CLINICAL TRIAL: NCT00001109
Title: Mononuclear Cell Phenotyping in Normal Children
Brief Title: A Blood Test to Look at Cells of the Immune System in Healthy Children
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: ACTG P1009; PACTG P1009
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2004-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Monocytes; Flow Cytometry; HIV Seronegativity; Phenotype; Lymphocyte Subsets
MeSH Terms: conditions — HIV Infections

SUMMARY:
The purpose of this study is to learn more about some of the immune cells in the blood (CD4 cells, for example) of healthy children in order to better understand the differences in the blood cells of children infected with HIV.

Because children's bodies are still developing, their cells are different from those of adults, and their bodies respond differently to infections such as HIV. In order to understand how immune cells grow and mature so that they can fight HIV, it is important to see how these cells behave in normal children.

DETAILED DESCRIPTION:
Early in life, the cells involved in immune selection differentiate into CD4+ and CD8+ cells. Currently there is insufficient information on the cell maturation and activation of these peripheral blood mononuclear cell (PBMC) subsets in normal children. The critical need for this information has been brought about by the pediatric HIV/AIDS epidemic, which requires the measurement of peripheral blood CD4+ T cells and other cells types for interpretation of HIV disease progression. The immunopathogenesis of pediatric HIV infection differs from that in adults but is not well understood. In order to better understand HIV disease progression in HIV-infected children, these PBMC subsets must be studied in normal children so that control values can be established.

Healthy infants, children, and adolescents presenting for routine care or elective surgery have a single blood sample obtained. Blood is used for complete blood count, peripheral blood mononuclear cell flow analysis for surface markers, and plasma and cell storage. Demographic information including age, sex, race, and ethnicity is obtained at the time of the blood draw. The reason for the patient's visit is also documented. No study drugs are administered or supplied as part of this study. Statistical analysis is used to estimate the median distribution of each CD4 and CD8 subset.

ELIGIBILITY:
Inclusion Criteria

A child may be eligible for this study if he/she:

* Is 0 - 18 years old.
* Is HIV-negative and is born to an HIV-negative mother.
* Is healthy (no serious infection or disease).
* Has signed informed consent of a parent or legal guardian if under 18.

Exclusion Criteria

A child will not be eligible for this study if he/she:

* Is pregnant or breast-feeding.
* Has already completed this study once before.
* Is taking prescription medications other than prescription vitamins.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 630

CONTACTS AND LOCATIONS:
Overall Officials: W Shearer, Study Chair; H Rosenblatt, Study Chair
Locations (45):
- United States (42):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Univ of South Alabama, Mobile, Alabama
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Cedars Sinai / UCLA Med Ctr, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Palm Beach County Health Dept, Riviera Beach, Florida
  - The Med Ctr Inc, Columbus, Georgia
  - Mt Sinai Hosp Med Ctr / Dept of Pediatrics, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Tulane Univ Hosp of New Orleans, New Orleans, Louisiana
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - UMDNJ - Robert Wood Johnson Med School / Pediatrics, New Brunswick, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Result] Shearer WT, Rosenblatt HM, Gelman RS, Oyomopito R, Plaeger S, Stiehm ER, Wara DW, Douglas SD, Luzuriaga K, McFarland EJ, Yogev R, Rathore MH, Levy W, Graham BL, Spector SA; Pediatric AIDS Clinical Trials Group. Lymphocyte subsets in healthy children from birth through 18 years of age: the Pediatric AIDS Clinical Trials Group P1009 study. J Allergy Clin Immunol. 2003 Nov;112(5):973-80. doi: 10.1016/j.jaci.2003.07.003. PMID 14610491